CLINICAL TRIAL: NCT07363356
Title: Drug Sensitivity Testing-Based Tumor Organoids to Guide Adjuvant Therapy After Hepatectomy for Primary Liver Cancer: A Prospective, Non-Randomized，Open-Label, Phase II Clinical Trial
Brief Title: Drug Sensitivity Testing-Based Tumor Organoids to Guide Adjuvant Therapy After Hepatectomy for Primary Liver Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, Shen Feng, Professor, Eastern Hepatobiliary Surgery Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EHBHKY2025-H030-P001
Record Dates: First submitted 2026-01-10; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma Resectable
Keywords: organoid;; drug-sensitive test;; adjuvant therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Organoid Drug Sensitivity Testing-Guided Therapy

INTERVENTIONS:
Drug: Organoid Drug Sensitivity Testing-Guided Therapy — Fresh tumor tissue from resection is used to establish and culture patient-derived organoids. Successful organoids undergo drug sensitivity testing against a predefined panel of drugs (Apatinib, Atezolizumab+Bevacizumab, Donafenib+Toripalimab, Sintilimab, FOLFOX). The most effective drug(s), based on IC50 and AUC values, are recommended for adjuvant therapy.

SUMMARY:
This is a single-center, prospective, non-randomized, open-label, phase II clinical trial aiming to evaluate the efficacy and feasibility of using patient-derived tumor organoid drug sensitivity testing (ODST) to guide personalized adjuvant therapy in patients with primary liver cancer (HCC) following curative liver resection. A total of 56 eligible patients will be enrolled. Tumor tissues obtained during surgery will be used to establish organoid cultures. Drug sensitivity testing will be performed on a panel of approved targeted and immunotherapeutic agents (including Apatinib, Atezolizumab + Bevacizumab, Donafenib + Toripalimab, Sintilimab, and FOLFOX) to identify the most effective treatment for each patient. Patients for whom organoid testing fails or results are unavailable within the specified timeframe will receive standard Lenvatinib treatment. The primary endpoint is Recurrence-Free Survival (RFS). Secondary endpoints include Overall Survival (OS) and safety profiles. The study seeks to provide a novel strategy for personalized adjuvant therapy in HCC to improve patient outcomes.

DETAILED DESCRIPTION:
1. Study Design:

   This is a single-center, prospective, non-randomized, open-label, phase II clinical trial conducted at the Third Affiliated Hospital of Naval Medical University. The study aims to validate the clinical utility of tumor organoid drug sensitivity testing in personalizing adjuvant therapy for hepatocellular carcinoma (HCC) after curative liver resection.
2. Study Population:

   The study will enroll 56 adult patients (aged 18-70) with primary HCC who have undergone curative liver resection and are at high risk of recurrence (e.g., tumor diameter >5 cm, multiple tumors, microvascular invasion, poor differentiation). Participants must have adequate organ function, an ECOG performance status of 0-1, and a life expectancy of >6 months.
3. Interventions:

   Organoid Drug Sensitivity Testing (ODST) Group: Fresh tumor tissue from resection is used to establish and culture patient-derived organoids. Successful organoids undergo drug sensitivity testing against a predefined panel of drugs (Apatinib, Atezolizumab+Bevacizumab, Donafenib+Toripalimab, Sintilimab, FOLFOX). The most effective drug(s), based on IC50 and AUC values, are recommended for adjuvant therapy.

   Control Group (Empirical Treatment): Patients for whom organoid construction fails, or valid drug sensitivity results are not available within 1 month, receive standard Lenvatinib treatment.
4. Study Endpoints:

   Primary Endpoint: Recurrence-Free Survival (RFS), defined as the time from treatment initiation to tumor recurrence.

   Secondary Endpoints:

   Overall Survival (OS)

   Safety and tolerability, assessed by the incidence and severity of adverse events (AEs, SAEs) according to NCI CTCAE v5.0.
5. Follow-up:

   Patients will be followed regularly with imaging (every 42±3 days initially, then every 3 months for the first year, and every 6 months thereafter) and laboratory assessments to monitor for recurrence and adverse events until death, withdrawal of consent, or study termination.
6. Statistical Analysis:

Sample size was calculated based on an assumed improvement in median RFS from 11.0 months (empirical group) to 33.0 months (ODST-guided group) (α=0.05, power=80%, 1:1 allocation, 10% dropout rate). Statistical analyses will be performed using SAS, with descriptive statistics for safety and efficacy analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 to 70 years.
2. Diagnosed with primary liver cancer according to the diagnostic criteria of the primary liver cancer (e.g., Guidelines for Diagnosis and Treatment of Primary Liver Cancer), with post-operative pathological confirmation of hepatocellular carcinoma (HCC). Patients must have at least one of the following high-risk pathological features: tumor diameter >5 cm, more than 3 tumors, presence of microvascular invasion, presence of minor macrovascular invasion, or poor pathological differentiation (Grade 3/4).
3. The subject or their legal guardian understands and voluntarily signs the informed consent form, and is willing and able to complete the scheduled visits, treatment plan, and laboratory tests as required by the protocol.
4. Life expectancy of more than 6 months.
5. No radiotherapy within 12 weeks prior to the first dose of study drug.
6. Liver function classified as Child-Pugh Class A or Class B with a score of 7.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Adequate organ and bone marrow function, defined as laboratory values meeting the following criteria within 7 days prior to randomization (without the support of blood transfusions, hematopoietic growth factors, albumin, or other corrective drugs within 14 days prior to obtaining the laboratory tests):

   8.1. Hematological:

   8.1. 2. Absolute Neutrophil Count (ANC) ≥1.5 × 10⁹/L

   8.1. 3. Platelet count (PLT) ≥75 × 10⁹/L

   8.1. 4. Hemoglobin (HGB) ≥9.0 g/dL

   8.2. Hepatic:

   8.2.1. Total Bilirubin (TBIL) ≤3 × Upper Limit of Normal (ULN)

   8.2.2. Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), and Alkaline Phosphatase (ALP) ≤5 × ULN

   8.2.3. Serum Albumin ≥28 g/L

   8.3. Renal:

   8.3.1. Serum Creatinine (Cr) ≤ 1.5 × ULN or Creatinine Clearance (CCr) ≥ 50 mL/min (calculated by Cockcroft-Gault formula)

   8.3.2. Urinalysis shows urine protein < 2+; if baseline urinalysis shows urine protein ≥ 2+, a 24-hour urine collection must demonstrate 24-hour urine protein quantification <1 g.

   8.4. Coagulation:

   8.4.1. International Normalized Ratio (INR) and Activated Partial Thromboplastin Time (APTT) ≤ 1.5 × ULN
9. For women of childbearing potential (WOCBP), a negative urine or serum pregnancy test must be confirmed within 3 days prior to receiving the first dose of study drug (Cycle 1, Day 1). If the urine pregnancy test is inconclusive, a serum pregnancy test is required. WOCBP and male subjects must agree to use adequate contraception during the observation period and for at least 8 weeks after the last dose of the study drug. A woman is considered not of childbearing potential if she is postmenopausal (≥1 year without menses) or has undergone surgical sterilization (bilateral oophorectomy, hysterectomy, or bilateral tubal ligation). Subjects (both male and female) with risk of pregnancy must use highly effective contraception (with a failure rate of <1% per year) during the entire treatment period and for 120 days after the last dose of study drug (or 180 days after the last dose of chemotherapy agents).

Exclusion Criteria:

1. Uncorrectable coagulopathy or significant bleeding tendency.
2. Evidence of any concurrent malignant disease.
3. Diagnosed with another malignancy within 3 years prior to the first dose, except for radically treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or carcinoma in situ that has undergone curative resection.
4. Requiring long-term anticoagulant or antiplatelet therapy that cannot be discontinued.
5. Presence of hepatic encephalopathy or refractory pleural effusion/ascites requiring therapeutic intervention.
6. Received other anti-tumor or systemic therapies within 2 weeks prior to enrollment, including:

   6.1. Chinese herbal medicines with clear anti-tumor properties.

   6.2. Chinese herbal medicines with anti-tumor indications or drugs with immunomodulatory effects (including thymosin, interferon, interleukin, except for local use to control pleural effusion).
7. History of systemic treatment for active autoimmune disease or ongoing immunosuppressive therapy:

   7.1. autoimmune disease requiring systemic treatment (e.g., disease-modifying agents, corticosteroids, or immunosuppressants) within 2 years prior to the first dose. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement) is not considered a form of systemic treatment.

   7.2. Systemic corticosteroid therapy (excluding topical, nasal, inhaled, or other non-systemic routes) or any other form of immunosuppressive therapy within 7 days prior to the first study dose. The use of physiologic doses of corticosteroids (≤10 mg/day prednisone or equivalent) is permitted.
8. Severe hepatic or renal insufficiency.
9. Presence of any severe or uncontrolled systemic disease, including but not limited to:

   9.1. Clinically significant, poorly controlled resting ECG abnormalities (e.g., complete left bundle branch block, second-degree or higher atrioventricular block, ventricular arrhythmias, or atrial fibrillation).

   9.2. Unstable angina, congestive heart failure (New York Heart Association (NYHA) Class ≥ II).

   9.3. Myocardial infarction within 6 months prior to randomization.

   9.4. History of esophageal or gastric variceal bleeding within 6 months prior to enrollment.

   9.5. Poorly controlled hypertension (systolic blood pressure >140 mmHg and/or diastolic blood pressure >90 mmHg).

   9.6. History of non-infectious pneumonitis requiring corticosteroid treatment within 1 year prior to the first dose, or current clinically active interstitial lung disease.

   9.7. Active tuberculosis.

   9.8. Active or uncontrolled infection requiring systemic therapy.

   9.9. Clinically active diverticulitis, intra-abdominal abscess, or gastrointestinal obstruction.

   9.10. Decompensated liver disease, acute or chronic active hepatitis.

   9.11. Unstable or active peptic ulcer disease, or patients with gastrointestinal bleeding.

   9.12. Poorly controlled diabetes mellitus (fasting blood glucose >10 mmol/L).

   9.13. Urinalysis showing urine protein ≥ ++ and confirmed 24-hour urine protein >1.0 g.

   9.14. Uncontrolled hypercalcemia (>1.5 mmol/L ionized calcium, or calcium >12 mg/dL, or corrected serum calcium > ULN), or symptomatic hypercalcemia requiring continued bisphosphonate therapy.

   9.15. Non-healing wound(s) or fracture(s).

   9.16. Psychiatric disorder that compromises the ability to comply with the treatment protocol.
10. Female subjects who are breastfeeding or pregnant.
11. Assessed by the investigator as being unable or unwilling to comply with the requirements of the study protocol.
12. Known allergy to any of the study drug(s) used in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free Survial(RFS) | Up to approximately 5 years
1year-RFS rate | 1-years
3years-RFS Rate | 3-years
5years-RFS Rate | 5-years

SECONDARY OUTCOMES:
Overall Survival（OS） | Up to approximately 5 years
Incidence of Adverse Events (AEs) | Up to approximately 4 years
  An adverse event is any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product.
1year-OS rate | 1-year
3years-OS Rate | 3-years
5years-OS Rate | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Feng Shen, Principal Investigator — Eastern Hepatobiliary Surgery Hospital
Locations (1):
- the Third Affiliated Hospital of Naval Medical University, Shanghai, Shanghai 200433/201805, Shanghai, China

IPD SHARING:
Plan to Share IPD: No